CLINICAL TRIAL: NCT03875677
Title: Using Neuroimage and Computational Modeling to Customize High-definition Transcranial Direct Current Stimulation Protocols for Facilitating Hand Function Recovery After Stroke
Brief Title: High-definition Transcranial Direct Current Stimulation for Facilitating Hand Function Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Chairman and Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017.155
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HD-tDCS group (Experimental): Constant current (1mA) will be applied for 20min and the anode will be placed over the defined target area
  Interventions: Device: HD-tDCS group
- Conventional tDCS group (Experimental): Constant current (1mA) will be applied for 20min and the anode will be placed over the standard C3/C4 position
  Interventions: Device: Conventional tDCS group
- Sham HD-tDCS group (Sham Comparator): The stimulator will be shut down after 30s of stimulation. The patients will feel the initial itching sensation at the beginning in order to evaluate the placebo effect.
  Interventions: Device: Sham HD-tDCS group

INTERVENTIONS:
Device: HD-tDCS group — 5 sintered Ag/AgCl ring electrodes will be used at a radius of ~5cm. The electrodes will be placed inside plastic electrode holders which will be filled with gel to have better contact with the scalp.
  Arms: HD-tDCS group
Device: Conventional tDCS group — A pair of 25 cm2 rubber electrodes enclosed in saline-soaked sponges and affixed to the head with rubber bands.
  Arms: Conventional tDCS group
Device: Sham HD-tDCS group — A pair of 25 cm2 rubber electrodes enclosed in saline-soaked sponges and affixed to the head with rubber bands.
  Arms: Sham HD-tDCS group

SUMMARY:
Transcranial direct current stimulation (tDCS) had recently been shown having feasibility in modulating cortical excitability transiently during motor training in a noninvasive way. The findings support that tDCS and motor practice can positively promote post-stroke motor learning to improve upper-limb motor recovery after stroke. A randomized controlled trial will be conducted with three groups: HD-tDCS, conventional tDCS and sham HD-tDCS. A 10-session training will be provided to evaluate the effectiveness of transient modulation of cortical excitability through tDCS with clinical assessment scores.

ELIGIBILITY:
Inclusion Criteria:

1. Hemiparesis subsequent to first-ever unilateral stroke for more than 6 months;
2. MCP and PIP finger joints can be extended to 180° passively;
3. Sufficient cognition to follow the experimental instructions

Exclusion Criteria:

1. Severe hand spasticity or hand deformity;
2. History of alcohol or drug abuse or epilepsy;
3. Bilateral brain infarcts;
4. Severe cognitive deficits;
5. Comprehensive aphasia;
6. Contraindications to tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | 3-month after the 10th session training
  The ARAT has total 19 items, divided into 4 categories (grasp, grip, pinch, and gross arm movement). It ranges from 3 to 0 (best to worse).

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (Upper Extremity) | 3-month after the 10th session training
  The maximum score is 66, divided into 33 items in the form of a 3-point scale (0-2), 0 is cannot perform and 2 performs fully.
Wolf Motor Function Test (WMFT) | 3-month after the 10th session training
  The WMFT measures upper limb ability through timed and functional tasks. It has 17 items, ranging from 0 to 5 (worse to best).
Magnetic Resonance Imaging | Baseline
  Functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No